CLINICAL TRIAL: NCT01113892
Title: Comparison of Safety and Primary Patency Between FUSION Vascular Graft With Bioline and EXXCEL Soft ePTFE (FINEST)
Brief Title: Study Comparing Synthetic Vascular Grafts in Patients With Peripheral Artery Disease (PAD) Who Require Artery Bypass.
Acronym: FINEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCV00001506
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Vascular Grafting

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized, single-blind (subject), parallel group, multicenter study in subjects with peripheral arterial occlusive disease (PAOD) who were scheduled to undergo femoral popliteal peripheral bypass surgery. Eligible subjects were randomly assigned in a 1:1 ratio to receive either FUSION Bioline or EXXCEL vascular graft.
Who Masked: Participant
Masking Description: This was a single-blind study. The surgeon and study site staff knew which vascular graft each subject received, but the subject did not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EXXCEL Soft (Active Comparator): A vascular graft comprised of extruded, expanded polytetrafluroethylene (ePTFE), indicated for use as a vascular prosthesis for replacement or bypass of diseased peripheral arteries (510(k) K962433).
  Interventions: Device: vascular grafts
- FUSION Bioline (Experimental): A synthetic vascular graft constructed of two layers. The inner layer is comprised of extruded, ePTFE. The outer layer is comprised of knit polyester textile. These two layers are fused together with a proprietary polycarbonate-urethane adhesive. The vascular graft also has a heparin coating on the graft's luminal surface. The Bioline coating is a bioactive surface coating consisting of a covalent Heparin Sodium coupled to immobilized recombinant human albumin.
  Interventions: Device: vascular grafts

INTERVENTIONS:
Device: vascular grafts — All devices will be used to treat patients with peripheral arterial occlusive disease

SUMMARY:
To demonstrate the patency and safety of vascular grafts: EXXCEL and FUSION Bioline.

DETAILED DESCRIPTION:
The study is a prospective, randomized, single-blind, two-arm, parallel group, multi-center study to evaluate the safety and efficacy of FUSION™ Vascular Graft with Bioline (heparin) coating, compared with EXXCEL Soft ePTFE in a peripheral bypass setting, to support a claim of substantial equivalence.

ELIGIBILITY:
Inclusion Criteria:

* Patient required either above-knee or below-knee femoral popliteal bypass;
* Patient had Category 1, 2, 3 4 or 5 chronic limb ischemia as defined by the Rutherford Categories - chronic limb ischemia severity classification scale.
* Patient was at least 21 years of age;
* Patient had postoperative life expectancy of >18 months;
* Patient was willing and able to have follow-up visits and examinations;
* Patient would not participate in other clinical trials that would conflict with this protocol
* Patient was willing and able to provide written, informed consent.

Exclusion Criteria:

* Patient had a previous history of bypass in the diseased extremity (below the iliacs arteries);
* Patient had percutaneous transluminal angioplasty or stenting of the target femoral or popliteal artery at the anticipated site of the proximal or distal anastomosis within the previous 30 days;
* Patient had active infection in the region of graft placement;
* Patient had an acute arterial occlusion requiring an emergent intervention;
* Patient needed a cardiac surgical procedure or a different vascular surgical procedure within 30 days of planned lower extremity revascularization. Planned endovascular procedures to address proximal stenotic lesions at the time of the index femoropopliteal bypass did not exclude a patient from the study;
* Patient required sequential extremity revascularizations or other procedures that require use of additional vascular grafts;
* Patient had known hypersensitivity or contraindication to aspirin;
* Patient had known coagulation disorders including hypercoagulability;
* Patient had previous instance of heparin-induced thrombocytopenia type 2 or has known hypersensitivity to heparin; Patient was currently treated with Coumadin (warfarin) that had not been stopped within 72 hours of the planned procedure
* Patient had severe chronic renal insufficiency (plasma/serum creatinine > 2.5 mg/dl), is undergoing hemodialysis.
* Patient had prior renal transplant;
* Patient had a stroke or myocardial infarction within 6 weeks of the procedure or had evidence of prior massive stroke (Modified Rankin Scale 3 or above);
* Patient had a myocardial infarction within 6 weeks prior to the procedure or had unstable angina pectoris;
* Patient had documented acute or suspected systemic infection;
* Patient was a woman of reproductive potential.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2012-12-18 (Actual); Study Completion 2013-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lumsden, MD, Principal Investigator — The Methodist Hospital Research Institute; Nicholas J. Morrissey, MD, Principal Investigator — NY Presbyterian-Columbia U Medical Center
Locations (25):
- United States (18):
  - University of Alabama-Birmingham Medical Center, Birmingham, Alabama
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - VA Palo Alto HCS, Palo Alto, California
  - University of South Florida - Tampa General, Tampa, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth- Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - NYU School of Medicine, New York, New York
  - NY Presbyterian Hospital - Columbia Univ Medical Center, New York, New York
  - Montefiore Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Dallas VA Medical Center, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Central Texas Veterans Health System, Temple, Texas
  - Scott & White, Temple, Texas
  - Norfolk Sentara - Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
- Czechia (6):
  - Fakulti Nemocnice Brno, Brno
  - Fakultni Nemocnice u sv Anny v Brno, Brno
  - University Hospital Plzen, Pilsen
  - Vseobecna Fakultni Nemocnice (VFN) Praha, Prague
  - IKEM Praha, Prague
  - Nemocnice Na Homolce, Prague
- Klinikum Karlsruhe, Karlsruhe, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lumsden AB, Morrissey NJ; Comparison of Safety and Primary Patency Between the FUSION BIOLINE Heparin-Coated Vascular Graft and EXXCEL Soft ePTFE (FINEST) Trial Co-investigators. Randomized controlled trial comparing the safety and efficacy between the FUSION BIOLINE heparin-coated vascular graft and the standard expanded polytetrafluoroethylene graft for femoropopliteal bypass. J Vasc Surg. 2015 Mar;61(3):703-12.e1. doi: 10.1016/j.jvs.2014.10.008. PMID 25720929
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from May 2010 to June 2012 at 18 sites in the United States (US) and 7 sites outside the US.
Pre-assignment Details: Subjects (209) were randomly assigned to FUSION Bioline (108) or EXXCEL (101) - 2 subjects in the FUSION Bioline group did not undergo surgery and are excluded from all analysis. One (1) of 207 treated subjects was included in efficacy analysis but excluded from safety analysis due to wrong treatment (FUSION instead of FUSION Bioline implanted).
Groups:
- EXXCEL Soft: Patients who were enrolled and treated with the EXXCEL Soft vascular graft.
- FUSION Bioline: Patients who were enrolled and treated with the FUSION Bioline vascular graft.
Period: Overall Study
Arm/Group | EXXCEL Soft | FUSION Bioline
Started | 101 | 106
Completed | 87 | 90
Not Completed | 14 | 16
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 2 | 4
Not completed — Graft no longer evaluable | 9 | 9

BASELINE CHARACTERISTICS:
Population: Of the 207 subjects treated, 203 were included in the efficacy analysis population. Four subjects were excluded due to data being unavailable for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | EXXCEL Soft | FUSION Bioline | Total
Number analyzed (Participants) | 100 | 103 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 43 | 102
  >=65 years | 41 | 60 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.76) | 65.7 (8.57) | 64.7 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 72 | 73 | 145
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 92 | 98 | 190
  African American | 8 | 2 | 10
  Hispanic | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 67
  Czechia | 64 | 63 | 127
  Germany | 4 | 5 | 9
Weight [Mean (Standard Deviation); unit: kg] | 83.1 (16.96) | 81.4 (17.06) | 82.2 (16.99)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index calculation based upon weight (in kg) divided by the height (in meters) squared.
  kg/m^2 | 27.8 (4.85) | 27.7 (4.86) | 27.7 (4.85)
Height [Mean (Standard Deviation); unit: cm] | 172.5 (8.1) | 171.2 (10.2) | 171.8 (9.2)
Rutherford Category [Count of Participants; unit: Participants]
  1-3 (claudication) | 76 | 71 | 147
  4-5 (limb threat) | 24 | 32 | 56
Ankle Brachial Index (ABI) [Mean (Standard Deviation); unit: Ratio] — The ankle brachial index (ABI) is the ratio between the systolic pressure measured at the ankle and the systolic pressure measured in the arm.
  Ratio | 0.56 (0.21) | 0.55 (0.24) | 0.55 (0.22)
Baseline medications [Count of Participants; unit: Participants]
  Aspirin | 85 | 87 | 172
  Clopidogrel | 15 | 13 | 28
  Any antiplatelet | 4 | 8 | 12
  Warfarin | 4 | 3 | 7
  Statin | 62 | 67 | 129
  Angiotensin-converting enzyme (ACE) inhibitor | 91 | 81 | 172
Comorbidities [Count of Participants; unit: Participants]
  Previous target limb intervention | 29 | 22 | 51
  Hyperlipidemia/hypercholesterolemia | 72 | 71 | 143
  Hypertension | 90 | 84 | 174
  Coronary artery disease | 35 | 38 | 73
  Obesity | 27 | 25 | 52
  Chronic obstructive lung disease | 16 | 24 | 40
  Cerebrovascular event | 12 | 7 | 19
  Liver disease | 7 | 6 | 13
  Bleeding disorder | 0 | 2 | 2
  Renal failure/dysfunction | 3 | 8 | 11
  Diabetes mellitus | 34 | 38 | 72
  Previous myocardial infarction | 22 | 21 | 43
  Arrhythmia | 8 | 11 | 19
  Congestive heart failure | 4 | 6 | 10
  Varicose veins | 17 | 20 | 37
Tobacco use [Count of Participants; unit: Participants]
  Current smoker | 51 | 54 | 105
  Prior smoker | 32 | 31 | 63
  Non-smoker | 17 | 18 | 35
Graft diameter [Count of Participants; unit: Participants]
  6 mm | 49 | 48 | 97
  8 mm | 51 | 55 | 106
Leg treated [Count of Participants; unit: Participants]
  Right | 47 | 50 | 97
  Left | 53 | 53 | 106
Site of proximal anastomosis [Count of Participants; unit: Participants]
  External iliac | 2 | 2 | 4
  Common femoral | 94 | 99 | 193
  Profunda femoral | 1 | 0 | 1
  Superficial femoral | 2 | 2 | 4
  Other | 1 | 0 | 1
Site of distal anastomosis [Count of Participants; unit: Participants]
  Above knee | 86 | 88 | 174
  Below knee | 14 | 14 | 28
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Patency
Description: A graft was considered to have primary patency if it had remained continuously patent (i.e., had continued blood flow through it) from the time of implantation and it had uninterrupted patency with no procedure performed on it, nor a procedure to address disease progression in the adjacent native vessel. Stenosis developing within the graft without remediation or occlusion was not considered a loss of primary patency. Assessed by duplex ultrasound imaging and ankle brachial index (ABI).
Time Frame: 6 months
Population: Subset of the efficacy analysis population with available data for analysis. The efficacy analysis population included all randomized subjects who met a study endpoint at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 100 | 103
Participants | 70 | 89
Statistical Analysis 1: Comparison: EXXCEL Soft vs FUSION Bioline; It was calculated that 200 participants randomized in a 1:1 fashion would have at least 80% power to detect a difference of 15% in the number of participants with primary patency between FUSION Bioline and EXXCEL groups at 6 months. It was assumed that the ratio of Above-Knee to Below-Knee procedures was 60:40; based on this, the primary patency rate for the combined Above-Knee and Below-Knee patients was 79%. Assumptions included a 10% withdrawal rate prior to the 6-month evaluation; Test type: Non-Inferiority — The non-inferiority margin was 15%. The following null hypothesis (H0) and alternative hypothesis (HA) were tested, with the primary patency rate at 6 months for FUSION Bioline (PF), and the primary patency rate at 6 months for EXXCEL (PE). H0: PF - PE < - 0.15; HA: PF - PE > - 0.15 An exact 1-sided test was used for the observed difference of patency rates between the FUSION Bioline (test) and EXXCEL (control) products; p < .0001, Exact 1-sided test — The threshold for significance was p = .05; Mean Difference (Net) = 16.4, 95% CI 2-sided [2.7 to 29.9] — Difference = Patency (Fusion Bioline) - Patency (EXXCEL)

2. Primary Outcome: The Number of Participants Meeting Composite Endpoint of Major Adverse Limb Events (MALE) and Periprocedural Death (POD)
Description: The composite endpoint included any of the following:
  * Major amputation - amputation that resulted in limb shortening (e.g., proximal to, but not including transmetatarsal amputations);
  * Major graft reintervention - placement of a new bypass graft at the same anatomic site, a jump/interposition graft, graft thrombectomy, graft excision, or graft thrombolysis;
  * Procedure-related death - any death within 30 days of the index procedure or within 30 days of any remedial procedure performed at the same anatomic site or as a result of the index procedure.
Time Frame: 6 months
Population: Safety population, defined as all randomized subjects who received the FUSION Bioline or EXXCEL vascular graft, analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 101 | 105
Participants
  Major amputation | 2 | 5
  Major graft reintervention | 31 | 17
  Procedure-related death | 1 | 1
  Any MALE or POD | 31 | 18
Statistical Analysis 1: Comparison: EXXCEL Soft vs FUSION Bioline; The number and percentage of subjects with a MALE or POD event were summarized by treatment group; Test type: Equivalence — Fisher's Exact test was used to evaluate whether subjects with any MALE event or POD were homogeneous across the treatment arms; p = .033, Fisher Exact

3. Secondary Outcome: Number of Participants With Primary Assisted Patency
Description: Primary assisted patency was defined as continued patency without thrombosis, with or without an endovascular or open surgical intervention to remediate a stenosis or other disorder of the graft.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 100 | 103
Participants | 73 | 89
Statistical Analysis 1: Comparison: EXXCEL Soft vs FUSION Bioline; Test type: Other; p = .017, Chi-squared; Proportion of subjects who achieved primary assisted patency for both treatment groups were compared using a Chi-Square test

4. Secondary Outcome: Number of Participants With Secondary Patency
Description: Secondary patency was defined as patency after some form of intervention to restore and maintain blood flow after occlusion.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 99 | 103
Participants | 80 | 91
Statistical Analysis 1: Comparison: EXXCEL Soft vs FUSION Bioline; Test type: Other; p = .137, Chi-squared; Proportion of subjects who achieve secondary patency for both treatment groups will be compared using a Chi-Square test

5. Secondary Outcome: Time to Hemostasis of Suture Hole Bleeding (Min)
Description: Time from the release of clamps until hemostasis, where hemostasis is defined as the absence of detectable bleeding from any of the suture holes.
Time Frame: Post-procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 100 | 102
minutes | 11 (10.63) | 3.5 (4.72)
Statistical Analysis 1: Comparison: EXXCEL Soft; Difference between groups were compared with the Wilcoxon Rank Sum Test; Test type: Other; p < .0001, Wilcoxon (Mann-Whitney)

6. Other Pre Specified Outcome: Number of Participants With Primary Patency
Description: A graft was considered to have primary patency if it had remained continuously patent (i.e., had continued blood flow through it) from the time of implantation and it had uninterrupted patency with no procedure performed on it, nor a procedure to address disease progression in the adjacent native vessel. Stenosis developing within the graft without remediation or occlusion was not considered a loss of primary patency.
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 99 | 101
Participants | 87 | 96

7. Other Pre Specified Outcome: Number of Participants With Primary Patency
Description: as for outcome 6
Time Frame: 12 months
Population: Subset of the efficacy analysis population with available data for analysis. The efficacy analysis population included all randomized subjects who met a study endpoint at 6 months. The 12 month efficacy analysis population for the 12 month results included those subjects who met the study endpoint at both 6 and 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 97 | 98
Participants | 65 | 75
Statistical Analysis 1: Comparison: EXXCEL Soft vs FUSION Bioline; Test type: Non-Inferiority — Repeated 6 month analyses for 12 month results.The non-inferiority margin was 15%. The following null hypothesis (H0) and alternative hypothesis (HA) were tested, with the primary patency rate for FUSION Bioline (PF), and the primary patency rate for EXXCEL (PE). H0: PF - PE < - 0.15; HA: PF - PE > - 0.15 An exact 1-sided test was used for the observed difference of patency rates between the FUSION Bioline (test) and EXXCEL (control) products, with a p-value ≤ .05 indicating significance; p = .0001, Exact 1-sided test; Mean Difference (Net) = 9.5, 95% CI 2-sided [-4.8 to 23.0]

8. Other Pre Specified Outcome: Number of Participants With Primary Assisted Patency
Description: as for outcome 3
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 99 | 101
Participants | 87 | 96

9. Other Pre Specified Outcome: Number of Participants With Primary Assisted Patency
Description: as for outcome 3
Time Frame: 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 97 | 98
Participants | 67 | 76
Statistical Analysis 1: Comparison: EXXCEL Soft vs FUSION Bioline; Test type: Other; p = .181, Chi-squared; Proportion of subjects who achieve primary assisted patency for both treatment groups will be compared using a Chi-Square test

10. Other Pre Specified Outcome: Number of Participants With Secondary Patency
Description: as for outcome 4
Time Frame: 30 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 99 | 101
Participants | 92 | 97

11. Other Pre Specified Outcome: Number of Participants With Secondary Patency
Description: as for outcome 4
Time Frame: 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | EXXCEL Soft | FUSION Bioline
Number analyzed (Participants) | 95 | 96
Participants | 77 | 80
Statistical Analysis 1: Comparison: EXXCEL Soft vs FUSION Bioline; Test type: Other; p = .68, Chi-squared; Proportion of subjects who achieve secondary patency for both treatment groups will be compared using a Chi Square test

ADVERSE EVENTS:
Time Frame: One Year
Description: An adverse event was defined as any side effect associated with the treatment procedure or device that produced an untoward medical effect or that had adverse health implications for the subject receiving the treatment. Adverse event data were collected from the time of procedure start through the last follow-up visit. Note that one (1) of 207 treated subjects was included in efficacy analysis but excluded from safety analysis due to wrong treatment (FUSION instead of FUSION Bioline implanted).
Groups:
- EXXCEL Soft: Patients who were enrolled and treated with the EXXCEL Soft vascular graft. The safety population was defined as all randomized subjects who received the FUSION Bioline or EXXCEL vascular graft, analyzed according to the treatment they received.
- FUSION Bioline: Patients who were enrolled and treated with the FUSION Bioline vascular graft. The safety population was defined as all randomized subjects who received the FUSION Bioline or EXXCEL vascular graft, analyzed according to the treatment they received. Note that one patient was randomized to the Fusion Bioline group but received the FUSION graft in error.
Arm/Group | EXXCEL Soft | FUSION Bioline
All-Cause Mortality (participants affected / at risk) | 2/101 | 4/105
Serious Adverse Events (participants affected / at risk) | 50/101 | 44/105
Other Adverse Events (participants affected / at risk) | 14/101 | 24/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXXCEL Soft (N=101) | FUSION Bioline (N=105)
Vascular graft thrombosis / Vascular graft occlusion (Injury, poisoning and procedural complications) | 32 (50) | 24 (34)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 3 (3) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Graft infection (Infections and infestations) | 0 (0) | 3 (3)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 3 (3) | 4 (4)
Peripheral ischaemia (Vascular disorders) | 4 (4) | 3 (3)
Femoral arterial stenosis (Vascular disorders) | 2 (2) | 0 (0)
Arterial stenosis limb (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Implant site effusion (General disorders) | 4 (4) | 3 (3)
Impaired healing (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Hernia obstructive (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Arterial bypass operation (Surgical and medical procedures) | 2 (2) | 0 (0)
Foot amputation (Surgical and medical procedures) | 0 (0) | 2 (2)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Debridement (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 2 (2) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXXCEL Soft (N=101) | FUSION Bioline (N=105)
Anaemia postoperative (Injury, poisoning and procedural complications) | 6 (6) | 11 (12)
Oedema peripheral (General disorders) | 9 (9) | 11 (11)
Impaired healing (General disorders) | 2 (2) | 6 (6)

LIMITATIONS AND CAVEATS:
Follow-up period was limited to 12 months. The inner layer is identical to EXXCEL, but FUSION Bioline also has an external polyester layer in addition to the heparin coating. Choices in perioperative care (surgeon discretion) may have differed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication or presentation of the results from a single site was not allowed until the preparation and publication of the multi-center results. Individual sites could publish or present information, provided that a draft was given to the sponsor for review and comment for a period that is at least 60 days prior to the first date of submission to allow the sponsor to review its content for accuracy, confidential information or patentable inventions.